CLINICAL TRIAL: NCT05679778
Title: PCO2 Gab as a Marker of Tissue Adequacy of Cardiac Output in Sever Shock State, Compared to Other Tissue Perfusion Indicators.
Brief Title: PCO2 Gab Marker of Tissue Adequacy of Cardiac Output in Shock State
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Muhammad Abd Elghany, MMAELGHANY, Assiut University
Other Study IDs: PCO2 gab in shock state
Record Dates: First submitted 2022-12-24; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Shock
Keywords: Delta PCO2 gap; Echocardiography; Left ventricle outflow tract velocity
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To assess validity of of central and pulmonary veno - arterial CO2 gradient to predict fluid responsiveness and to guide fluid management and determine the cut off point to continue or stop resuscitation.
2. comparison between PCO2 gab and left ventricular outflow tract velocity time integral to determine whether to continue or stop resuscitation and whether PCO2 gab is a surrogate of cardiac output or not.

DETAILED DESCRIPTION:
Assessing the adequacy of oxygen delivery with oxygen requirements is one of the key-goal of hemodynamic resuscitation. Clinical examination, lactate and central or mixed venous oxygen saturation (SvO2 an ScvO2 respectively) all have their limitations (Gavelli et al., 2019). The veno- arterial difference in CO2 tension (delta CO2 or PCO2 gap) is not indicator of anaerobic metabolism since it is influenced by the oxygen consumption. By contrast, it reliably indicates whether blood flow to remove is sufficient to carry CO2 from prepheral tissues to the lung in view of its clearance: it, thus, reflects the adequacy of cardiac output with the metabolic condition (valley et al., 2013). The gap is a marker of adequacy of venous blood flow to remove CO2 produced rather than a marker of tissue hypoxia (Vallet et al., 2013).

The gab can be calculated from simultaneous sampling of central venous blood from a central vein catheter and arterial blood.

Determining the delta PCO2 during resuscitation of septic shock Patients might be useful when deciding when to continue resuscitation despite a central venous oxygen saturation>70% associated with elevated blood lactate levels. because a high blood lactate level is not a discriminatory factor in determining the source of that stress, an increased delta PCO2 (>6 mmHg) could be used to identify Patients who still remain inadequately resuscitated.

Fluid responsiveness in shocked patients is conventionally defined as an increase of at least 10% to 15% in stroke volume in response to a fluid challenge. Assessment of response to a fluid challenge can be guided with echocardiography. It is achieved by measuring left ventricular outflow tract velocity time integral (LVOT VI) immediately before and after fluid challenge (miller et al; 2016).

ELIGIBILITY:
Inclusion Criteria:

* all critical ill-patients with acute physiological assessment and chronic health evaluation II score (APACHE II score)≥25 with central line insertion, in the critical care uint of internal medicine department of Assuit university hospital in the period between January 2023 to January 2024.

Exclusion Criteria:

1. Pateints with poor echocardiographic window.
2. Pateints with APACHE II score < 25.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All critical ill-patients of all age groups, who presented shocked, with good echocardiographic window, with CVC insertion.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of heamodynamic state, need of fluid resuscitation and inotropes. | January 2023 to January 2024
  Assessing need of fluid resuscitation and need of inotropes to continue resuscitation to maintain stable heamodynamic status.

SECONDARY OUTCOMES:
Duration of hospital stay, time to control various clinical and laboratory abnormalities (BP, PP, RR, lactate, renal chemistry) and development of complications as; pulmonary edema and use of mechanical ventilation. | January 2023 to January 2024
  Use of delta PCO2 in assessing of hemodynamic stability to shortcut hospital stay, time to control clinical and laboratory abnormalities and decrease the possibility of development of complications as pulmonary edema and use of mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Ali, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gavelli F, Teboul JL, Monnet X. How can CO2-derived indices guide resuscitation in critically ill patients? J Thorac Dis. 2019 Jul;11(Suppl 11):S1528-S1537. doi: 10.21037/jtd.2019.07.10. PMID 31388457